CLINICAL TRIAL: NCT02256865
Title: Hormonal Mechanisms of Sleep Restriction
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Peter y. Liu, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 30068-01
Record Dates: First submitted 2014-09-22; First posted 2014-10-06 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Insulin Resistance
Keywords: Sleep Restriction; Insulin Resistance; Testosterone; Cortisol
MeSH Terms: conditions — Insulin Resistance | interventions — Ketoconazole; Hydrocortisone; Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo and Drug Group 2 (Placebo Comparator): Placebo pills and gel is used in place. Placebo for Ketoconazole is taken 4 times a day Placebo for Hydrocortisone is taken 3 times a day Placebo for testosterone gel is applied once a day.
  Interventions: Drug: Ketoconazole; Drug: Hydrocortisone; Drug: Testosterone; Drug: Placebo for ketoconazole; Drug: Placebo for hydrocortisone; Drug: Placebo for testosterone
- Drug and Placebo Group 1 (Active Comparator): Ketoconazole is taken 4 times a day Hydrocortisone is taken 3 times a day Testosterone gel is applied once a day
  Interventions: Drug: Ketoconazole; Drug: Hydrocortisone; Drug: Testosterone; Drug: Placebo for ketoconazole; Drug: Placebo for hydrocortisone; Drug: Placebo for testosterone

INTERVENTIONS:
Drug: Ketoconazole — Ketoconazole is taken 4 times a day
  Other Names: Nizoral
Drug: Hydrocortisone — Hydrocortisone is taken 3 times a day
  Other Names: Cortef, Cortril, Hydrocortone
Drug: Testosterone — Testosterone gel is applied once a day
  Other Names: AndroGel
Drug: Placebo for ketoconazole — Placebo for ketoconazole
Drug: Placebo for hydrocortisone — Placebo for hydrocortisone
Drug: Placebo for testosterone — Placebo for testosterone

SUMMARY:
The purpose of this study is to study the effects of sleep restriction on the production of two hormones, cortisol and testosterone. The investigators aim to show that changing these hormones leads to insulin resistance, which is an important cause of type 2 diabetes mellitus. The investigators may also study the effect of sleep restriction on your food intake and cravings, mood, inflammation, metabolism (including bone), and other hormones. Inflammation is your body's response to stress and injury. Bone metabolism is a process of how your body regenerates (renews) new bone cells and removes old bone cells. Hormones are natural substances (materials) that are produced in the body and that influences (effects) the way the body grows or develops.

DETAILED DESCRIPTION:
Screening Visits

* To see if you are able to take part in this study, you will first have an outpatient visit at the CTRC (Clinical and Translational Research Center). This visit will take about 90 minutes.
* The following tests/procedures will be done at this visit:

  * We will ask you about your medical history and past health
  * We will give you a physical examination (including digital rectal examination of the prostate gland if you are over the age of 40)
  * We will ask you to answer sleep, mood and general health screening questionnaires.
  * We will ask you to complete a questionnaire to help us understand how testosterone and other hormones control sexual function and drive.
  * We will draw about 1 tablespoon of blood from a needle placed in a vein in your arm for routine safety tests and to check to see if you have any hormonal problems.
  * We will give you an ECG (recording of heartbeat). For this test we will attach 12-lead sensors to your chest.
  * We will collect urine sample from you for a drug screening test.
  * A dietitian will review meal plans for the inpatient stay (Study Visit 1 and 3 only).

If the first screening visit shows that you are able to continue to take part in this study, you will continue the screening part of the study at home. The following will be done at home: We will ask you to undergo an at-home actigraphy and keep a daily sleep diary for two weeks to document your sleeping habits. For the actigraphy you will be asked to wear a small wrist-watch like device. This device will monitor and record your motion, and will also test your sleep and wake periods. It may be worn for up to 2 weeks, 24 hours per day (except while taking a shower).

If the results of the at-home actigraphy show that you are still able to take part in this study, you will continue the final part of the screening procedure which is an inpatient visit to conduct a sleep study. The following tests/procedures will be done for this final screening visit: We will ask you to come into the sleep laboratory to sleep overnight (sleep study). A technician will attach the leads (wires) to your body and you will need to keep these leads on during the night. The attached wires will be connected to a machine to measure chest and abdominal (stomach area) movements, airflow at your mouth and lips, blood oxygen level, muscle tone, eye movements, heart rate and electrical activity of the brain. In the morning, the technician will remove the attached wires.

If the exams, tests and procedures during the screening visits show that you can continue to be in the study, you will have 2 inpatient visits and 2 outpatient clinical visits.

Before beginning the study, we will assign you to one of the two study groups described below. Which one you are assigned to will be decided by chance (like tossing a coin) and you will have a one in two chance of being in any one group. A computer program will place you in one of the study groups.

GROUP 1: If you are assigned to group 1, then you will receive active drug during visit 1 (first inpatient visit) and placebo (inactive drug which is same as receiving no drug) during visit 3 (second inpatient visit). GROUP 2: If you are assigned to group 2, then you will receive placebo (inactive drug which is same as receiving no drug) during visit 1 (first inpatient visit) and active drug for visit 3 (second inpatient visit).

Neither you nor your study doctor can choose the group you will be in. Neither your study doctor or his staff nor you will know which study group or medicine you will be receiving. However should a medical emergency occur, this information will be made immediately available to your study doctor.

During the inpatient visit when you receive active drug, you will receive: Ketoconazole pills. You will swallow these pills every 6 hours (4 times per day). Testosterone gel. You will rub this gel into your skin once a day in the morning. Hydrocortisone pills. You will swallow these pills 3 times a day.

During the inpatient visit when you receive placebo (inactive drug), you will receive:

* Inactive placebo pills (looks like ketoconazole). You will swallow these pills every 6 hours (4 times per day).
* Inactive placebo gel (looks like testosterone gel). You will rub this gel into your skin once a day in the morning.
* Inactive placebo pills (looks like hydrocortisone). You will swallow these pills 3 times a day.

Night before First Inpatient Visit Before coming to the CTRC for your first inpatient visit, you will be asked to sleep 10 hours for two consecutive nights (from 10 PM to 8 AM) at home. During your sleep, you will be wearing an actiwatch to monitor your sleep at home. You cannot drink any alcohol during this 2 day period. We will send you a text message or telephone you to remind you to sleep during these times and not to drink alcohol. The inpatient study visit will be cancelled if you didn't have enough sleep at home or if you consumed alcohol.

Study Visit 1 (First Inpatient) For this visit we will ask you to arrive at the CTRC no later than 5 PM on the first day. We will allow you to go home sometime after lunch after the 5th night. We will give you breakfast, lunch and dinner at set times while you are in the CTRC. The meals are standard, so that what you may have eaten before will not interfere with the study results. The following tests/procedures will be done at this visit: We will download the information from your actiwatch to verify your sleep at home. We will be putting external leads on your body, as occurred during the sleep study, so that we can continuously check your sleep EEG, actiwatch activity and heart rate. We will expose you to dim light (this is so we can measure your "body clock"). From 7 PM until your bedtime every night, saliva will be collected hourly so we can measure your "body clock". We will ask you to fill out a short questionnaire to measure how sleepy you are, how hungry you are and do a computerized test of cognitive function every 2 hours (on odd, not even, hours). This will take about 5 minutes. Starting at 8PM on your first night, urine will collected until 8AM of the following day. This will be repeated every 12-hour period whilst in-lab for measurements of components of in the urine. We will give you an Oral Glucose Tolerance Test (OGTT) in the morning of the first and last days (on two occasions) while you are in the CTRC. The OGTT is the test that measures the body's ability to use a type of sugar, called glucose, which is the body's main source of energy.

* Before the test begins, we will insert a cannula into a vein in your arm and a sample of blood will be taken. The cannula is a small plastic tube through which we will sample your blood. It is inserted over a metal needle into your vein. The metal needle is removed once the cannula is in place.
* We will ask you to drink a liquid that is high in glucose (75 grams).
* In the first hour, we will draw about 5ml (1 teaspoon) of blood will be taken from the cannula every 5 minutes.
* In the second hour, about 5ml (1 teaspoon) of blood will be taken from the cannula every 10 minutes
* In the third hour, about 5ml (1teaspoon) of blood will be taken from the cannula every 20 minutes.
* We will draw an additional 10ml (2 teaspoons) of blood to measure inflammation, hormones, gene expression, and bone metabolism
* The entire test will take about 3 hours.

We will give you an opportunity to sleep before we discharge you and we will test you for sleepiness. Arrangements will be made for you to be driven home if necessary. During this time you cannot drink caffeinated drinks, or use nicotine products.

Study Visit 2 (First Outpatient) This visit will take place one week after you are discharged from your first inpatient visit. At this visit we will ask you about any side effects and draw about 1 tablespoon of blood for complete blood count and routine chemistry check, including liver function tests.

Study Visit 3 (Second Inpatient) This visit will take place one week after your first outpatient visit (about 2 weeks after your first inpatient visit). This visit is identical the first inpatient study Visit 1. For this visit, if you received active study drug during your first inpatient visit, you will receive a placebo. If you received the placebo during the first inpatient study Visit 1, then you will receive active study drug during this visit.

Study Visit 4 (Second Outpatient) This visit will take place one week after you are discharged from your second inpatient visit. At this visit we will ask you about any side effects and draw about 1 tablespoon of blood for complete blood count and routine chemistry check, including liver function tests.

All visits A total of about half a pint (16 tablespoons) of blood will be collected for this study. We will collect less than what you would donate to the blood bank.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 22-45 years
* Willingness to provide written informed consent
* Stable weight over preceding 6 weeks
* Body Mass index (BMI) 20-28 kg/m2

Exclusion Criteria:

* Unable or unwilling to provide IRB-approved informed consent
* Clinical disorders and/or illnesses
* Current medical or drug treatment, as assessed by questionnaire
* History of brain injury or of learning disability
* Vision or hearing impairment unless corrected back to normal
* Anemia (Hct <38%)
* History of psychiatric illness
* Clinically significant abnormalities in blood and urine, and free of traces of drugs Other endocrine abnormalities including hypothyroidism or adrenal failure; primary gonadal disease as indicated by serum LH or FSH concentration >10 or >15 IU/L, respectively, hyperprolactinemia indicated by prolactin >25ug/L
* Type 2 Diabetes (HgbA1C)
* Current smoker
* Recent or concurrent drug or alcohol abuse
* Blood donation in previous eight weeks
* Travel across time zones within one month of entering the study
* Sleep or circadian disorder
* Shift work within three months of entering the study
* Irregular bedtimes (not between 6 and 10 hours in duration)
* Unoperated obstructive uropathy, recurrent prostatitis, indeterminate prostatic nodularity, Hx or Suspicion of cancer of the prostate gland or PSA >4ng/ml
* Previous adverse reaction to sleep deprivation or any of the drugs to be administered
* Concurrent participation in another research study

Ages: 22 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2017-11 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 3 years
  Insulin sensitivity determined by minimal model of a frequently sampled oral glucose tolerance test (OGTT).This method is extensively validated, and previously utilized by us.

SECONDARY OUTCOMES:
Disposition index | 3 years
  Disposition index (determined by minimal model of the same OGTT)
C-peptide glucose dose-response | 3 years
  C-peptide glucose dose-response (also calculated from the same OGTT)
Lapses on Psychomotor Vigilance Task | 3 years
  Measure of psychomotor performance
Karolinska Sleepiness Scale | 3 years
  Measures sleepiness
Urinary Catecholamines | 3 years
  Measures sympathetic/parasympathetic activity
Heart Rate Variability | 3 years
  Measures sympathetic/parasympathetic activity
Free Fatty Acid Concentrations | 3 years
  Measures potential mediator of insulin resistance
Inflammatory marker panel | 3 years
  blood interleukin-6, sTNFr2, IL1ra, CRP, NFkB concentrations
Computerized cognitive testing | 3 years
  Two card gambling task, modified Sternberg working memory task
Bone turnover panel | 3 years
  P1NP (bone formation marker) and NTX (bone resorption marker)
Food cravings, | 3 years
  Food Craving Index
Assessment of mood states. | 3 years
  Profile of Mood States (POMS)
Food intake | 3 years
  meal and snack consumption calculation
Hunger measurement | 3 years
  Flint visual analogue scale

OTHER OUTCOMES:
Epigenetics | 3 years
  Explorative study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Y Liu, MD PhD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles Biomedical Research Institute, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Byrne NA, Yuen F, Niaz W, Liu PY. Sleep and the Testis. Curr Opin Endocr Metab Res. 2021 Jun;18:83-93. doi: 10.1016/j.coemr.2021.03.002. Epub 2021 Mar 11. PMID 33937581
- [Background] O'Byrne NA, Yuen F, Butt WZ, Liu PY. Sleep and Circadian Regulation of Cortisol: A Short Review. Curr Opin Endocr Metab Res. 2021 Jun;18:178-186. doi: 10.1016/j.coemr.2021.03.011. Epub 2021 May 5. PMID 35128146
- [Result] Liu PY, Lawrence-Sidebottom D, Piotrowska K, Zhang W, Iranmanesh A, Auchus RJ, Veldhuis JD, Van Dongen HPA. Clamping Cortisol and Testosterone Mitigates the Development of Insulin Resistance during Sleep Restriction in Men. J Clin Endocrinol Metab. 2021 Aug 18;106(9):e3436-e3448. doi: 10.1210/clinem/dgab375. PMID 34043794
- [Derived] Zhang W, Piotrowska K, Chavoshan B, Wallace J, Liu PY. Sleep Duration Is Associated With Testis Size in Healthy Young Men. J Clin Sleep Med. 2018 Oct 15;14(10):1757-1764. doi: 10.5664/jcsm.7390. PMID 30353813
- Available data/document: Statistical Analysis Plan — https://research.labiomed.org/redcap/redcap_v7.2.2/FileRepository/file_download.php?pid=174&id=19887 — Data Analysis Plan available by request to PI